CLINICAL TRIAL: NCT04513795
Title: EARLY-MYO-SEPSIS (EARLY Assessment of MYOcardial Injury in Sepsis Patient) Registry
Brief Title: EARLY-MYO-SEPSIS Registry
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EARLY-MYO-SEPSIS
Record Dates: First submitted 2020-08-10; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The diagnosis and pathophysiology of sepsis-induced cardiac dysfunction remain unknown. This registry is to evaluate characteristics of sepsis patients by multi-modalities imaging, including echocardiography, cardiovascular magnetic resonance imaging in 300 patients in 5 sites. Subjects will be followed up to 2 years.

DETAILED DESCRIPTION:
Approximately 20-30 million patients worldwide suffer from sepsis every year, which is increasing at the rate of 8% to 13% per year. It is possible that sepsis progress to multiple organ dysfunction in the early stage, with a fatality of 30% to 60%. Myocardium is one of the most vulnerable tissue under the abnormal 'inflammation storm'.Cardiac dysfunction is one of the important predictors for mortality of sepsis.Patients with myocardial depression have an apparently higher mortality rate (70%) as compared with septic patients without cardiac impairment (20%).

Although several trials had explored the diagnosis and treatment of sepsis-induced cardiac dysfunction, the effective characteristic depict and effective therapy remain incompletely understand.

This is a prospective, multi-center, non-randomized, observational registry study of sepsis patients that undergo multi-modality imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patiants meets the criteria of Sepsis 3.0 as below:
* Sepsis is a lifethreatening organ dysfunction caused by a dysregulated host response to infection
* 1 patients in ICU：
* 1.1 have at least one organ dysfunction
* 1.2 SOFA score ≥2
* 2 patients not in ICU
* 2.1 have at least one organ dysfunction
* 2.2 SOFA score or qSOFA score ≥2

Exclusion Criteria:

* 1. Patient who is unable to comply with the follow-up schedule.
* 2. Patient who has any medical conditions that in the opinion of the investigators will not be appropriate to participate in the study.
* 3. Patient has a life expectancy of less than 6 months due to any condition

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients were diagnosed as sepsis or suspected as sepsis
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
composite of death, stroke, heart failure | 2 years
  composite of death, stroke, heart failure

SECONDARY OUTCOMES:
day of hospitalization | through study completion, 2 months
  day from admission to discharge